CLINICAL TRIAL: NCT07279532
Title: Clinical Study of Adjuvant Surufatinib Therapy for Postoperative High-risk Neuroendocrine Tumors Based on the Ninth Edition of the AJCC Staging System
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1173
Record Dates: First submitted 2025-11-24; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Neuroendocrine Neoplasms (Tumours)
MeSH Terms: conditions — Neoplasms | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Surufatinib 200mg, administered orally once daily (QD), for 6 months as postoperative adjuvant therapy.
  Interventions: Drug: surufatinib

INTERVENTIONS:
Drug: surufatinib — Surufatinib 200mg, administered orally once daily (QD), for 6 months as postoperative adjuvant therapy.

SUMMARY:
The following issues warrant in-depth investigation: further refinement of staging by primary tumor site, the increasing prognostic weight of T classification, risk assessment for lymph node metastasis and postoperative recurrence/distant metastasis, and whether NET G3 with poor prognosis requires more aggressive postoperative intervention. This study plans to enroll patients classified as Stage III according to the AJCC 9th Edition staging system, including NET G1/G2 and all G3 patients, for a clinical trial on postoperative adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent and voluntarily participate in the study.
2. Aged 18-80 years, male or female.
3. Confirmed as Stage III NET G1/G2 or any-stage NET G3 after surgical treatment.
4. Other postoperative NET patients deemed by the investigator to have high-risk factors.
5. Adequate organ function meeting the following criteria (no use of any blood components, cell growth factors, or corrective drugs within 14 days prior to the first dose of the study drug): (i) Absolute Neutrophil Count (ANC) ≥1.5×10⁹/L; (ii) Platelets ≥100×10⁹/L; (iii) Hemoglobin ≥8 g/dL; (iv) Total Bilirubin ≤1.5 × ULN; ALT and AST ≤2.5 × ULN (or ≤5 × ULN if liver metastases are present); (v) Serum Creatinine ≤1.5 × ULN or Creatinine Clearance >60 mL/min (Cockcroft-Gault formula).
6. Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours before the first study drug dose and use effective contraception during the study and for at least 3 months after the last dose. Male subjects with female partners of childbearing potential must use effective contraception during the study and for 3 months after the last dose.

Exclusion Criteria:

1. Major surgery, open biopsy, or significant trauma within 28 days prior to the first dose.
2. History of severe or poorly controlled interstitial lung disease.
3. Poorly controlled hypertension (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg) despite antihypertensive medication.
4. Poorly controlled cardiovascular diseases, including but not limited to:

   (i)NYHA Class II or higher heart failure; (ii) Unstable angina; (iii) Myocardial infarction within the past year; (iv) Clinically significant supraventricular or ventricular arrhythmias poorly controlled with or without intervention.
5. Significant bleeding tendency or clinically significant bleeding within 3 months prior to the first dose (e.g., gastrointestinal bleeding, hemorrhagic gastric ulcer, vasculitis).
6. Arterial/venous thrombotic events within 6 months prior to the first dose (e.g., transient ischemic attack, cerebral hemorrhage, cerebral infarction, deep vein thrombosis, pulmonary embolism). Superficial vein thrombosis may be enrolled if deemed eligible by the investigator.
7. Concurrent active malignancy requiring treatment, except for adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix.
8. Pregnancy or lactation.
9. Any other condition deemed by the investigator to potentially lead to study discontinuation (e.g., severe comorbid illnesses, abnormal laboratory values, psychosocial issues).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival（RFS） | 4 years
  Refers to the time from when a patient achieves complete response after anticancer therapy or surgery until the occurrence of disease recurrence or death from any cause.

SECONDARY OUTCOMES:
Overall Survival （OS） | 4 years
  Refers to the time from the start of randomization (or the start of treatment in a single-arm trial) until death due to any cause.
Adverse Event (AE) | 4 years
  In a drug clinical trial, it refers to all adverse medical events that occur in subjects after receiving the investigational medicinal product, which can manifest as symptoms, signs, diseases, or laboratory abnormalities, but are not necessarily causally related to the investigational medicinal product.

OTHER OUTCOMES:
Biomarkers | 4 years
  Concentrations of NSE and ProGRP in blood samples, evaluated as percentage changes at each tumor assessment from baseline to treatment